CLINICAL TRIAL: NCT05086263
Title: Effects of Virtual Reality MRI Preparedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey I Gold, PhD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHLA-21-00107
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Educational Problems
Keywords: Virtual Reality; Magnetic resonance imaging; Radiology
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A schedule of randomization matching and stratified in age and gender will be computer generated and used to determine which group the child will be placed in. Neither the investigator nor child will know which group they are in until after the parent and child complete the first set of questionnaires
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No VR) Randomization (No Intervention): Participants would take the same questionnaires as the VR interventional group except the RT questionnaire. Then they will proceed with their MRI.
- VR Randomization (Experimental): The virtual reality MRI training will be conducted immediately after completion of the questionnaires in a distraction free room. The training explains the procedure to the viewer and addresses common questions that individuals often have regarding an MRI. Using audio/visual cues and biofeedback training is aimed to mimic the experience of the MRI with real audio recordings of image acquisition, in order to adequately train the view to stay still in an MRI procedure. The research subject will continue with their regularly scheduled MRI. The modified Yale Preoperative Anxiety Scale (mYPAS) is an observational measure and will be completed by research staff.
  Interventions: Device: Pico G2 4k

INTERVENTIONS:
Device: Pico G2 4k — On this virtual reality headset, it will be loaded with an educational virtual reality mock MRI training titled "Ready Teddy". This training explains the procedure to the viewer and addresses common questions that individuals often have regarding an MRI. Furthermore, using audio/visual cues, when the viewer moves their head too much in a MRI like setting they are reminded to stay still. Biofeedback training is aimed to mimic the experience of the MRI with real audio recordings of image acquisition, in order to adequately train the view to stay still in an MRI procedure.
  Arms: VR Randomization

SUMMARY:
Magnetic resonance imaging is an important and increasingly prevalent imaging modality used in healthcare. Children often find the procedure anxiety provoking causing difficulty in staying still and providing quality images. The use of preparation techniques including play therapy and role play utilizing such tools as a fiberglass mock MRI have shown to reduce anxiety and facilitate better image quality. Modalities of preparation including Virtual Reality (VR) pose as an alternative to habituate children for a MRI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages of 8-9 years inclusive
* Child scheduled for a clinical MRI at CHLA.

Exclusion Criteria:

* Child is younger than 8 years or older than 9 years. These are the bottom end of age ranges that are frequently sedated.
* Children who have metal in their bodies that cannot participant in an MRI.
* Medical history that may affect brain development that may confound ability to complete an MRI without sedation.
* Children suffering from epilepsy or history of seizures who may react poorly to a virtual reality intervention.
* Child who has a history of MRI acquisition where habituation and preparedness may not be needed.
* Child with English as a second language due to restrictions of research team.
* Child with implantable medical devices or personal medical devices that may be affected by the study device's radio waves

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Childhood Anxiety Sensitivity Index (CASI) | Approximately 5 minutes to one hour before procedure
  This 18-item measure utilizes a three-point Likert scale (none (1), some (2), a lot (3)) to assess how negatively patients view anxiety symptoms. Items are summed with a higher score indicating greater anxiety sensitivity.
Number of Participants with Successful Imaging without Sedation | Up to thirty minutes after intervention
  A successful image will be produced after MRI. Failure would mean the child is rescheduled for another MRI with sedation.
Visual Analogue Scale (VAS) | Approximately 5 minutes to one hour before intervention
  The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children
Faces Pain Scale-Revised (FPS-R) | Approximately 5 minutes to one hour before procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Child Anxiety Meter State (CAM-S) | Approximately 5 minutes to one hour before procedure
  The child is asked to color a thermometer that has ten marks to indicate their level of anxiety they feel at the moment. The meter can be translated to a 0-10 scale with higher score indicating greater anxiety.
Child Anxiety Meter Trait (CAM-T) | Approximately 5 minutes to one hour before procedure
  The child is asked to color a thermometer that has ten marks to indicate their level of anxiety they usually feel at home. The meter can be translated to a 0-10 scale with higher score indicating greater anxiety.

SECONDARY OUTCOMES:
Demographics | Up to one hour before intervention
  24 Item questionnaire which asks parents demographic questions regarding socioeconomic data.

OTHER OUTCOMES:
Satisfaction Questionnaire | Immediately after intervention
  45 item questionnaire using a four point scale (strongly agree, agree, disagree, and strongly disagree) to gauge ease of use and satisfaction using the VR headset. Higher scores reflect greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Gold, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bharti B, Malhi P, Khandelwal N. MRI Customized Play Therapy in Children Reduces the Need for Sedation--A Randomized Controlled Trial. Indian J Pediatr. 2016 Mar;83(3):209-13. doi: 10.1007/s12098-015-1917-x. Epub 2015 Oct 19. PMID 26477350
- [Background] Carter AJ, Greer ML, Gray SE, Ware RS. Mock MRI: reducing the need for anaesthesia in children. Pediatr Radiol. 2010 Aug;40(8):1368-74. doi: 10.1007/s00247-010-1554-5. Epub 2010 Feb 26. PMID 20186541
- [Background] Eatough EM, Shirtcliff EA, Hanson JL, Pollak SD. Hormonal reactivity to MRI scanning in adolescents. Psychoneuroendocrinology. 2009 Sep;34(8):1242-6. doi: 10.1016/j.psyneuen.2009.03.006. Epub 2009 Apr 5. PMID 19346079
- [Background] Power JD, Mitra A, Laumann TO, Snyder AZ, Schlaggar BL, Petersen SE. Methods to detect, characterize, and remove motion artifact in resting state fMRI. Neuroimage. 2014 Jan 1;84:320-41. doi: 10.1016/j.neuroimage.2013.08.048. Epub 2013 Aug 29. PMID 23994314
- See also: Related Info — http://readyteddy.io